CLINICAL TRIAL: NCT04265248
Title: Effectiveness of Cervical Exercises Using Virtual Reality Headsets on Pain and Disability in Patients With Chronic Neck Pain
Brief Title: Evaluation of the Effects of Virtual Reality in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josue Fernandez Carnero (Other)
Collaborators: CEU San Pablo University (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: URJC-02/2020
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain; Pain, Neck
Keywords: Virtual reality; Chronic pain; Neck pain; Physiotherapy; Exercise
MeSH Terms: conditions — Chronic Pain; Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The subjects will use "Fulldive VR" as the first degree of difficulty where only tilt movements are necessary, for the second degree of difficulty the game "VR Ocean Aquarium 3D" will be used, where bending, extension and rotation movements will be integrated, also introducing a sensory element to integrate the sound of the sea.
  For these patients to perform the same work as group 2, the physiotherapist will have to count and control in each exercise the number of movements that the patient performs so as not to exceed the proposed dose in the active comparator group (3 sets of 10 repetitions of each exercise).
  Interventions: Device: Virtual Reality Headset
- Exercise (Active Comparator): The subjects perform the exercises provided by the researchers. Which consist of neck exercises in all ranges of movement (inclinations and rotations to both sides), apart from flexion and extension.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Device: Virtual Reality Headset — The subjects will wear the Virtual Reality Headset with a mobile phone inserted into it with the applications Full Dive VR and VR Ocean Aquarium 3D.
  Arms: Virtual Reality
Behavioral: Exercise — The subjects will perform evidence-based exercises for the neck.
  Arms: Exercise

SUMMARY:
The main objective of this research is to assess the effectiveness of virtual reality as a treatment to reduce pain and disability in patients with chronic neck pain compared to a regular exercise program for the neck.

DETAILED DESCRIPTION:
Chronic neck pain is one of the most common causes of pain and disability. Its prevalence is approximately 15% in adults and it is one of the main causes of medical leave and the increase of drug consumption. Recent research has found that neck pain is a common pathology among the population. Among the variables associated with neck pain, besides rheumatology, include genetic, psychopathological variables (such as depression, anxiety, coping skills, somatization), sleep disorders, smoking and a sedentary lifestyle, among others. All those variables alter the nervous system in a proprioceptive level, so that deep and superficial flexor, as well as the rest of the muscles, they do not receive correct information that prevents them from processing properly the obtained information. Therefore, alterations also occur at central nervous system levels as in the processing of pain and its control by inhibitory descending systems.

One of the most effective treatments for this pathology is active exercise. The main objective is the activation and strengthening of the deep flexor muscles by craniocervical flexion. It is also important to re-educate all the movements performed with the neck; extension, rotation and inclination are essential movements that also require good initial control of deep flexor muscles and its dynamism is essential to interact with our surroundings.

The action observation which consists of observing an action carried out by another person is based on the ability of the nervous system to assimilate the images seen and process them until they reach the motor cortex, and thanks to the mirror neurons, the painful pattern decreases until it disappears. Thus, visualising a painful situation provokes and evokes in the brain, a painful experience, even when this is not actually happening. Therefore, it has been proved that it can produce changes in the motor cortex since the observation reinforces the cortical representation of the action, thus achieving an improvement in strength and functionality in patients with chronic pain.

Taking all this into account, in this study the investigators propose the idea of working with virtual reality headset in patients with chronic neck pain. This treatment offers great visual, auditory and vestibular feedback that makes it an attractive and stimulating exercise for the patient. It has the ability to individualize treatments and patient needs. These virtual environments can graduate and increase the complexity of the task while decreasing the help and feedback provided by the therapist. The goal of a virtual reality based treatment is to make patients more participatory in their real environments as independently as possible. It is an innovative treatment that does not demand a great financial cost for its use.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic chronic neck pain.
* Understands and accept the informed consent form.
* Meets the age limits criteria.

Exclusion Criteria:

* Patients under 18 or over 65 years old.
* Pregnancy.
* Specific neck pain due to metastases, neoplasms, infectious or inflammatory. processes, fractures, or traumatic history of cervical injury.
* Positive neurological signs or evidence of spinal cord compression (abnormal diffuse sensitivity, hyperreflexia or diffuse weakness).
* Cervical osteoarthritis.
* Polyarthrosis.
* Neck Pain associated with vertigo (vestibular involvement).
* Neck Pain associated with whiplash injuries.
* Previous cervical surgeries.
* Headaches before cervicalgia without cervical origin.
* Inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in cervical range of movement. | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  Measured with goniometer by the physiotherapists.
Changes in pain perception. | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  Self reported Visual Analog Scale. Minimum value is 0 (best); Maximun value is 10 (worst).
Changes in Neck Pain and Disability Perception | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  10 Neck Disability Index Scale that must be answered with a numeric value between 0 (no disability) and 5 (complete disability), with a maximum score of 50 points, with higher scores indicating greater neck disability.

SECONDARY OUTCOMES:
Changes in levels of Catastrophism. | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  13 item Pain Catastrophic Scale that must be answered with a numeric value between 0 (not at all) and 4 (all the time), with a maximum score of 52 points, with higher scores indicating greater pain catastrophizing.
Changes in Kinesiophobia, levels of fear to movement. | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  11 item Tampa Scale for Kinesiophobia, the final score can range between 11 and 44 points, with higher scores indicating greater perceived kinesiophobia.
Changes in Fear-avoidance behaviours. | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  Fear-avoidance Beliefs Questionnaire . The instrument consists of two subscales, a four-item physical activity subscale, and a seven-item work subscale. Each item is scored from 0 to 6 and summed to produce the subscale score. Possible scores range from 0-28 to 0-42, with higher scores indicating greater fear avoidance beliefs.
Changes in levels of hyperalgesia to pressure and maximum pressure tolerance. | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  Pressure Pain Thresholds using an algometer on first finger, trapezius muscle and tibia.
Changes in endogenous pain inhibition mechanisms. | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  Conditioned pain modulation and temporal summation (windup), using the algometer and an occlussion band.
Changes in Anxiety Related to Pain | Before and after the treatment (2 weeks), after 1 month and after 3 months.
  20 item Pain Anxiety Symptoms Scale scoring from 0 to 100 with higher scores indicating greater pain-related anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: David Morales Tejera, Msc., Phdc, Principal Investigator — Escuela Internacional de Doctorado de la Universidad Rey Juan Carlos
Locations (2):
- Spain (2):
  - Universidad Rey Juan Carlos, Alcorcón, Madrid
  - CEU San Pablo, Madrid, Madrid, Montepríncipe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de-la-Puente-Ranea L, Garcia-Calvo B, La Touche R, Fernandez-Carnero J, Gil-Martinez A. Influence of the actions observed on cervical motion in patients with chronic neck pain: a pilot study. J Exerc Rehabil. 2016 Aug 31;12(4):346-54. doi: 10.12965/jer.1632636.318. eCollection 2016 Aug. PMID 27656633
- [Background] Kim JY, Kwag KI. Clinical effects of deep cervical flexor muscle activation in patients with chronic neck pain. J Phys Ther Sci. 2016 Jan;28(1):269-73. doi: 10.1589/jpts.28.269. Epub 2016 Jan 30. PMID 26957772
- [Background] Borisut S, Vongsirinavarat M, Vachalathiti R, Sakulsriprasert P. Effects of strength and endurance training of superficial and deep neck muscles on muscle activities and pain levels of females with chronic neck pain. J Phys Ther Sci. 2013 Sep;25(9):1157-62. doi: 10.1589/jpts.25.1157. Epub 2013 Oct 20. PMID 24259936
- [Background] Gallego Izquierdo T, Pecos-Martin D, Lluch Girbes E, Plaza-Manzano G, Rodriguez Caldentey R, Mayor Melus R, Blanco Mariscal D, Falla D. Comparison of cranio-cervical flexion training versus cervical proprioception training in patients with chronic neck pain: A randomized controlled clinical trial. J Rehabil Med. 2016 Jan;48(1):48-55. doi: 10.2340/16501977-2034. PMID 26659920
- [Background] Sarig Bahat H, Weiss PL, Sprecher E, Krasovsky A, Laufer Y. Do neck kinematics correlate with pain intensity, neck disability or with fear of motion? Man Ther. 2014 Jun;19(3):252-8. doi: 10.1016/j.math.2013.10.006. Epub 2013 Nov 9. PMID 24291364
- [Background] Palacios-Cena D, Alonso-Blanco C, Hernandez-Barrera V, Carrasco-Garrido P, Jimenez-Garcia R, Fernandez-de-las-Penas C. Prevalence of neck and low back pain in community-dwelling adults in Spain: an updated population-based national study (2009/10-2011/12). Eur Spine J. 2015 Mar;24(3):482-92. doi: 10.1007/s00586-014-3567-5. Epub 2014 Sep 11. PMID 25208501
- [Background] Nederhand MJ, Ijzerman MJ, Hermens HJ, Turk DC, Zilvold G. Predictive value of fear avoidance in developing chronic neck pain disability: consequences for clinical decision making. Arch Phys Med Rehabil. 2004 Mar;85(3):496-501. doi: 10.1016/j.apmr.2003.06.019. PMID 15031840
- [Background] Rudolfsson T, Djupsjobacka M, Hager C, Bjorklund M. Effects of neck coordination exercise on sensorimotor function in chronic neck pain: a randomized controlled trial. J Rehabil Med. 2014 Oct;46(9):908-14. doi: 10.2340/16501977-1869. PMID 25182501
- [Background] Sarig Bahat H, Sprecher E, Sela I, Treleaven J. Neck motion kinematics: an inter-tester reliability study using an interactive neck VR assessment in asymptomatic individuals. Eur Spine J. 2016 Jul;25(7):2139-48. doi: 10.1007/s00586-016-4388-5. Epub 2016 Jan 30. PMID 26831536
- [Background] Sarig Bahat H, Takasaki H, Chen X, Bet-Or Y, Treleaven J. Cervical kinematic training with and without interactive VR training for chronic neck pain - a randomized clinical trial. Man Ther. 2015 Feb;20(1):68-78. doi: 10.1016/j.math.2014.06.008. Epub 2014 Jul 5. PMID 25066503